CLINICAL TRIAL: NCT04068298
Title: A Prospective, Single-center Study of Temperature Gradients for Sepsis Severity and Fluid Resuscitation
Brief Title: Temperature Gradients for Sepsis Severity and Fluid Resuscitation
Acronym: sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Zhongqing Chen, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: 2018cr047; 320.6750.18431 (Other Grant/Funding Number: Wu Jieping Fund)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Sepsis
Keywords: sepsis; temperature gradient; microcirculation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment and treatment of Septic Shock (SS) is a thorny issue in current care. Fluid resuscitation is one of the key measures for SS treatment. Current fluid resuscitation is dominated by empirical treatment or early target-directed therapy. The former has a clear goal of recovery, and the latter is complicated to implement and has many complications. It is known that patients with SS due to insufficient tissue perfusion, the distribution of blood flow in the peripheral center to the center, may lead to an increase in the central-peripheral-room temperature difference, suggesting that this index has potential value for direction of fluid resuscitation. This study intends to measure the severity of SS and efficacy of fluid resuscitation by measuring the "central-peripheral-room temperature" gradient of patients as well as comparing temperature gradient with hemodynamic indexes (PICCO) and indexes of ultrasound capacity assessment, providing more convenient indicators for sepsis and fluid resuscitation assessment.

DETAILED DESCRIPTION:
Sepsis remains a great challenge for clinicians. Early and timely fluid resuscitation is the basic measure for the treatment of sepsis. It is important to quickly diagnose the severity of sepsis and evaluate the effects of fluid resuscitation. Existing monitoring methods such as blood pressure, urine volume, blood lactate, central venous oxygen saturation (ScvO2), cardiac output (CO), stroke volume variability (SVV), etc. have certain limitations or invasive disadvantages. Clinically, effective and convenient non-invasive means are needed for monitoring. Present research revealed that microcirculatory dysfunction and tissue hypoperfusion have a very important role in the pathophysiological mechanism of sepsis, and will be associated with severe organ dysfunction, which is closely related to serious adverse prognosis. Importantly, tissue hypoperfusion can cause central and peripheral body temperature changes. Studies have shown that clinical assessment of peripheral skin temperature can identify potential severe organ dysfunction in patients with stable hemodynamics. The latest study found that patients with septic shock have greater central-peripheral body temperature differences than sepsis patients, and the temperature difference between peripheral-room temperature is smaller. That is, the central-peripheral-room temperature gradient changes show a reduction of tissue perfusion, suggesting microcirculatory disorders and organ dysfunction. In addition, the body temperature gradient is simple and non-invasive, and is a bedside indicator that predicts tissue perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years old.
* Patients with sepsis or septic shock who meet the diagnostic criteria for sepsis 3.0 and who are routinely treated according to 《Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016》.
* Get informed consent within 2 hours.

Exclusion Criteria:

* Age <18 years old.
* A confirmed pregnancy or urine pregnancy test is positive.
* Patients with septic shock at low temperature (central body temperature <35 °C).
* The informed consent of the legal representative of the subject was not obtained.
* Known liver disease affecting peripheral perfusion assessment, such as vascular occlusive vasculitis, multiple arteritis, and Raynaud's disease.
* Any disease that restricts the use of fluid resuscitation, such as: heart failure, major cardiac surgery, post-cardiopulmonary resuscitation, severe heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects were patients with sepsis and/or septic shock in the Department of Critical Care Medicine, Southern Hospital from September 2019 to September 2022.
Sampling Method: Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | three years
  Rate of all-caused mortality at 28 days

SECONDARY OUTCOMES:
ICU Length of stay | three years
  Days of participants stay in the intensive care unit (ICU)
Hospital Length of stay | three years
  Days of participants stay in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang hospital, Guangzhou, Guangdong, China